CLINICAL TRIAL: NCT00411021
Title: Endometrial Sampling (Pipelle)in IVF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-05-3674-MB-CTIL
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2006-12-13 (Estimated); Status verified 2006-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

INTERVENTIONS:
Procedure: Pipelle (Endometrial Sampling)

SUMMARY:
A prospective cross-over randomized study aimed to test the hypothesis that local injury of the endometrium increases the implantation rate in the successive cycle. Seventy IVF patients will be randomly selected to undergo either endometrial biopsies or minimal cervical scratch on days 8-10 and 21-23 of their cycle, preceding the IVF treatment. If not pregnant, the women will continue for another IVF cycle, preceded by endometrial or cervical scratch complimentary to their procedure in the first cycle. The main major outcomes will include pregnancy rate, implantation rate, endometrial thickness, abortion rate, live births and embryo quality.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF treatment
* Repeated Implantation failure

Exclusion Criteria:

* PID or suspected PID
* Undiagnosed Irregular Bleeding

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70

CONTACTS AND LOCATIONS:
Overall Officials: Micha Baum, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- IVF Unit, Sheba Medical Center, Ramat Gan, Israel